CLINICAL TRIAL: NCT04095676
Title: Intrapleural Fibrinolysis and DNase Versus VATS for the Treatment of Pleural Empyema: a Randomized, Controlled Trial
Brief Title: VATS Surgery Compared to Drainage in the Treatment of Pleural Empyema
Acronym: FIVERVATS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Decker Christensen (Other)
Collaborators: Odense University Hospital (Other); Rigshospitalet, Denmark (Other); Aalborg University Hospital (Other)
Responsible Party: Sponsor-Investigator, Thomas Decker Christensen, Consultant, Professor, MD, DMSc., Ph.D, Aarhus University Hospital
Organization: Aarhus University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FIVERVATS1
Record Dates: First submitted 2019-09-05; First posted 2019-09-19 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-08

CONDITIONS: Pleural Empyema
MeSH Terms: conditions — Empyema, Pleural | interventions — Drainage

STUDY DESIGN:
Intervention Model Description: * Randomized, controlled study
  * Not blinded (open label)
  * National multicenter study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- VATS / surgical group (Experimental): The VATS procedure must be completed as soon as possible and no later than 48 hours after randomisation. The surgery is performed with the patient in a 90 degree sideways position, using general anesthesia. Access is obtained through one to three ports, followed by purification and possibly decortication, and insertion of one pleural drain (sizes 24 - 32F) at the end of surgery. 20 ml Marcain is used as local analgetic and applied at the incision sites or as a nerve block. In the VATS group, suction on drain (- 15 cm H20) is applied in the first day after the procedure. Operator must have relevant training and competencies corresponding to the specialist level within the relevant specialty and be registered and approved by the steering committee.
  Interventions: Procedure: VATS group
- Drain and intrapleural therapy group (Active Comparator): Pigtail is applied as soon as possible and within 48 hours after randomisation. Drain placement is carried out using ULS. Operators (conductors of the procedure) must have relevant training and competencies corresponding to the specialist level within the relevant specialty and be approved by the steering committee to conduct the procedure. A pigtail catheter (minimum 10F) is inserted. Operator determines the size of drain and whether drain placement is done with one-step or Seldinger technic.
  The intrapleural therapy consists of treatment with the following two drugs:
  * intrapleural Actilyse® (alteplase) 10 mg twice daily for three days
  * intrapleural Pulmozyme® (DNase) 5 mg twice daily for three days
  Interventions: Procedure: Drain and intrapleural therapy group

INTERVENTIONS:
Procedure: VATS group — VATS procedure with drainage, including rinse with NaCl
  Arms: VATS / surgical group
Procedure: Drain and intrapleural therapy group — Drainage with pigtail and Intrapleural therapy
  Arms: Drain and intrapleural therapy group

SUMMARY:
Pleura empyema is a frequent disease with a high morbidity and a mortality rate of approximately 15%.

Pleura empyema is characterized by the passage of three stages (I - III). The aim of treating the disease is to remove the infection and provide fully expansion of the lung.

The initial treatment at the early stage of the disease (stage I) is simple drainage. In clinical practice, stages II and III are treated alike.

Current standard treatment for these stages is drainage with ultrasound (ULS) -guided pigtail. Simultaneously with drainage, an intrapleural fibrinolyticum can be given. A potential better alternative is surgery in terms of Video Assisted Thoracoscopic Surgery (VATS). The theoretical advantage of early surgery is that patients undergo rapid, definitive treatment. Furthermore, surgery can ensure optimal drain placement. How best to treat these patients (drainage or surgery) is still under clinical evaluation and depends to a great extent on local clinical practice. It is only to a limited extent based on scientific evidence.

The aim of this study is to determine if there is a difference in outcome in patients diagnosed with stage II and stage III empyema who either receive primary VATS surgery or ULS guided drainage and intrapleural therapy (fibrinolytic (altaplasm) with DNase (Pulmozyne ®)) The primary outcome is Hospitalization time and secondary outcomes is e.g. mortality, health related costs and quality of life.

The present study can thus provide new and highly relevant knowledge as well as change the treatment of these patients, both nationally and internationally.

It is planned that a total of 184 patients will be included in the project. The study takes place as a collaboration between all four thoracic surgical departments and the major pulmonary medicine departments in Denmark. In addition, the study has international collaborators/consultants who will provide counselling in connection with the study.

DETAILED DESCRIPTION:
Intrapleural Fibrinolysis and DNase versus VATS for the treatment of pleural empyema: a randomized, controlled trial

BACKGROUND

Pleural empyema is a disease with an infection inside the chest cavity, often as a result of a pneumonia. In Denmark there are approximately 500 new cases per year. Patients often have longer duration of hospitalization, and the disease carries a significant morbidity and mortality rate of approximately 15%. The state of pleura empyema is characterized by the passage of three stages (I - III):

* Parapneumonic effusion (stage I)
* Fibropurulent stage (stage II)
* Chronic organizing stage (stage III)

The aim of treating the disease is to remove the infection and provide fully expansion of the lung.

In our study we want to find the optimal method for treating patients in stage II and III.

The initial treatment at the early stage of the disease (stage I) is simple drainage and the disease at later stages can be treated with surgical intervention. In clinical practice, stages II and III are treated alike. Current standard treatment for these stages is drainage with ultrasound (ULS) -guided pigtail with a minimum size of 10 F. Simultaneously with drainage, an intrapleural fibrinolyticum can be given, but the indication and evidence for this is discussed. In the MIST II study, fibrinolytic (alteplase) was combined with DNase, and the authors found a positive effect using this combination.

Previously, surgery was associated with a significant morbidity and, to a lesser extent, mortality. The surgery was conducted as open surgery using a thoracotomy. Today, it can often be performed as a Video Assisted Thoracoscopic Surgery (VATS), which can be performed with a very low morbidity and mortality. It has been advocated that patients should be operated very early in the process, but the evidence is weak. In a Cochrane review on surgical versus non-surgical treatment of pleura empyema, two studies with adult patients have been included. None of the studies have a size or methodological quality that makes it possible to determine whether VATS should be included as part of the standard treatment of these patients. In children (aged <15 years), a randomized, controlled study of 50 patients in each group was conducted. It found no difference in outcome between fibrinolyticum and VATS, but no fixed treatment algorithm has been established for this age group. Furthermore, these results cannot be generalized to an adult population.

The theoretical advantage of early surgery is that patients undergo rapid, definitive treatment and surgery can ensure optimal drain placement. The potential advantages in early surgery are reduced mortality, admission time, and fewer late complications. In addition, it is estimated that an increased number of early-operable patients may reduce the proportion of patients, who will later be thoracotomized, as early surgery may be performed as VATS. However, there is the inherent risk of an operation and thereby the increased costs of the surgical procedure when compared to simple drainage. However, this could possibly be outweighed by reduced drug consumption, reduced need for supplemental drainage, shorter duration of admission, and reduced morbidity after discharge.

Accordingly, it is necessary to determine whether early VATS should be introduced as standard therapy in patients with fibropurulent stage (stage II) and the chronic organizing stage (stage III).

Hypothesis • Patients over 18 years with a fibropurulent stage (stage II) or a chronic organizing stage (stage III) pleural empyema will have a significantly reduced time of hospitalization, if they undergo a VATS operation compared to ULS-guided pigtail drainage and fibrinolyticum (Acitlyse® (altaplasm)) with DNase (Pulmozyne®)

Aim of study

• To determine the difference in outcome in patients diagnosed with complex parapneumonic effusion (stage II), and pleural empyema (stage III) who are treated either VATS surgery or TUS guided drainage and intrapleural therapy (fibrinolytic (Alteplase) with DNase (Pulmozyme®)) as first line treatment.

Expected improvements If this trial is positive for the primary and/or the secondary outcomes, it could potentially change and strengthen the treatment of patients with this disease, both nationally and internationally. We investigate both clinical parameters, patient satisfaction and economical aspects (cost-effectiveness) in relation to pleura empyema treatment, so it will cover many aspects of this disease. If the trial is neutral, it will provide valuable data on intervention that is currently commonly used for this disease and can guide the treating physician to choose the adequate treatment based on the local preferences.

METHODS Design

* Randomized, controlled study
* Not blinded (open label)
* National multicenter study

Inclusion and exclusion criteria

Inclusion criteria:

* 18 years or more on the day of hospitalization
* Must be able to provide informed consent
* Acute hospitalization within the last 48 hours
* Meeting diagnostic criteria for community acquired pleural infection using the following criteria:

  1. A clinical presentation compatible with pleural infection AND
  2. Has pleural fluid which is either:

     1. purulent pleural fluid or
     2. gram stain positive or
     3. culture positive or
     4. acidic with pH < 7.2 or
     5. low pleural fluid glucose (< 2 mmol/L) in the absence of accurate pH measurement or
     6. septated pleural fluid on ultrasound

Exclusion criteria:

* • Pregnancy. Prior to inclusion of fertile women (defined as the period from menarche to postmenopause) a negative pregnancy test must be available
* Breastfeeding
* Declared terminally ill or a predicted survival of less than 3 months
* Previous intrathoracic surgery (within <1 year on the same side of the thorax as where the parapneumonic effusion/pleural empyema is located
* Previously (within <1 year) hospitalized with with complex parapneumonic effusion (stage II) or pleural empyema (stage III)
* Drainage during the current admission on the same side of the thorax (excluding diagnostic pleural puncture)
* Hospitalization within 7 days prior to current hospitalization
* Previous allergic reaction to alteplase or DNase
* Use of alteplase therapy contraindicated:

  * Ongoing treatment with oral anticoagulant incl. new oral anticoagulants (e.g. warfarin (Marevan), Dabigatranetexilat (Pradaxa), Rivaroxaban (Xarelto), Apixaban (Eliquis), Endoxaban (Lixiana))
  * Significant ongoing bleeding or within last six months
  * Known haemorrhagic diathesis
  * Previous or suspected intracranial hemorrhage
  * Suspected subarachnoidal hemorrhage or condition following subarachnoidal hemorrhage from aneurysm
  * All forms of damage to the central nervous system (e.g. cerebral tumors, aneurysm, intracranial / spinal surgery)
  * Recent (within 10 days) cardiac resuscitation, birth, or perforation of non-compressible blood vessel (e.g. puncture of v. subclavia, v. jugularis)
  * Severe, uncontrolled arterial hypertension
  * Bacterial endocarditis, pericarditis
  * Acute pancreatitis
  * Documented ulcerative gastrointestinal disease within last 3 months, esophagal varices, arterial aneurysm, arterio-venous malformations
  * Tumor / malignancy with an increased risk of hemorrhage
  * Severe liver disease, including liver failure cirrhosis, portal hypertension (esophagal varices), and active hepatitis
  * Large operation or significant trauma within previous 3 months

Endpoints

Primary endpoint:

• Length of hospital stay, where admission time is defined as the time from first admission in the course of the hospitalization and to the completion of treatment defined as time of discharge from hospital without need of any additional invasive treatment.

Secondary endpoints:

* Hospitalization time when patients are stratified in subgroups (Stage, TUS score, RAPID score)
* Length of hospital stay after commencement of intervention
* Days at home up to 30 days after intervention (DAH30)
* 30-day and in-hospital mortality
* Time from randomization to commencement of intervention
* Drainage time measured in days
* Proportion of patients where primary intervention could be considered as definitive treatment
* Complications ranked by Clavien-Dindo classification and Comprehensive Complication Index (CCI)
* Need for additional thoracic surgery within 12 months after hospitalization
* Consumption of painkillers during hospitalization and within 12 months after hospitalization
* Lung physiology within 12 months after hospitalization
* Quality of life and patient reported outcomes within 12 months after hospitalization
* Health related costs within 12 months after hospitalization

Randomization

Patients will be randomized 1:1 to either:

1. VATS procedure with drainage
2. TUS-guided pigtail catheter placement and intrapleural therapy with Actilyse and DNase Block randomization with varying block size will be used to get an equal number of patients in both groups. There will be stratification for each surgical center in the randomization. The randomization is conducted via a REDCap (Research Electronic Data Capture), (REDCap Consortium, Vanderbilt University Medical Center, Tennessee, USA).

   Blinding Patients and responsible health care staff will not be blinded. Research staff not involved in the treatment of the included patients are blinded to treatment allocations until data analyses are complete. Assessment of different scoring systems (e.g. TUS and radiology score) are blinded to the extent that it is practically possible.

   Patient population and selection All patients admitted during the diagnosis of pleural empyema or pleural effusion without specification (diagnostic codes: DJ 86, DJ 86.1, DJ 86.9, DJ 90.9), Stages II and III will be potential candidates, whether they are hospitalized at a Regional Hospital or at a University Hospital.

   Practical issues regarding inclusion of patients Patients who immediately meet the criteria for inclusion and are interested in participating are informed by one of the project participants or project nurses from the thoracic surgery department or other relevant department where the patient is hospitalized. The physical location of information and randomization will vary with the local organization of hospitals and departments. If the patient is randomized to VATS, the patient is transferred to one of the four centers where there is a thoracic surgical department. If the patient is randomized to ULS guided drainage and intrapleural therapy, the patient is transferred to one of the specialized pulmonology departments participating in the project.

   Intervention Drain and intrapleural therapy group Pigtail is applied as soon as possible and within 48 hours after randomisation. Drain placement is carried out using ULS. Operators (conductors of the procedure) must have relevant training and competencies corresponding to the specialist level within the relevant specialty and be approved by the steering committee to conduct the procedure. A pigtail catheter (minimum 10F) is inserted. Operator determines the size of drain and whether drain placement is done with one-step or Seldinger technic.

   The intrapleural therapy consists of treatment with the following two drugs:
   * intrapleural Actilyse® (alteplase) 10 mg twice daily for three days
   * intrapleural Pulmozyme® (DNase) 5 mg twice daily for three days Both drugs are administered twice daiyly through the pigtail catheter and are left for one hour in the pleural cavity by blocking the drain (e.g. closing the three-way-stopcock / use of a pean forceps). The installation of the drugs in the pleural cavity is performed seperately with a time interval between administrations of at least two hours. Actilyse® (alteplase) is preparred by diluting 10 mg Actilyse® (alteplase) in the solvent liquid (10 ml) supplied alongside the drug in a 50 ml syringe. This mixture is further diluted by drawing isotonic NaCl into the syringe until the total volume of fluid in the syringe is 30 ml. Following this preparation the mixture is injected into the pleural cavity using the pigtail catheter. Pulmozyme® (DNase) is prepared by drawing 5 ml Pulmozyme® (DNase) (1mg/ml)(5 ml = 2 Pulmozyme cannisters) into a 50 ml syringe. This mixture is further diluted by drawing isotonic NaCl into the syringe until the total volume of fluid in the syringe is 30 ml. Following this preparation the mixture is injected into the pleural cavity using the pigtail catheter.

   VATS group The VATS procedure must be completed as soon as possible and no later than 48 hours after randomisation. The surgery is performed with the patient in a 90 degree sideways position, using general anesthesia. Access is obtained through one to three ports, followed by purification and possibly decortication, and insertion of one pleural drain (sizes 24 - 32F) at the end of surgery. 20 ml Marcain is used as local analgetic and applied at the incision sites or as a nerve block. In the VATS group, suction on drain (- 15 cm H20) is applied in the first day after the procedure. Operator must have relevant training and competencies corresponding to the specialist level within the relevant specialty and be registered and approved by the steering committee.

   After the procedure Randomized patients are transferred to a specialized respiratory medical department or remain at the thoracic surgical department.

   Saline flushes In both groups following completion of the intervention flushes of 30 ml normal saline will be given three times daily to ensure tube patency.

   Antibiotics

   The empiric antibiotic treatment used in all centers is in accordance with the national guidelines from the Danish Society for Cardiothoracic Surgery and Danish Society for Respiratory Medicine [19, 20]. Treatment is initiated as intravenous treatment. Type of antibiotic treatment can be subsequently adjusted depending on results of microbiological tests. Change to oral treatment can be done when all of the following three criteria are met:
   * Clinical improvement of the patient (e.g. no fever/fever, improved general condition)
   * Paraclinically satisfactory response (with respect to decreases in leukocytes and CRP's)
   * Drain/pigtail is removed This means that 14 days i.v. treatment will not be given as standard. The duration of i.v. antibiotic treatment will therefore be individual based on the application of the above criteria. The overall duration of treatment of antibiotic is 6 weeks as standard.

   Other treatments and supportive care

   All patients are:
   * Offered specialized lung physiotherapy
   * Screened for and given additional nutritional support
   * Treated with painkillers in accordance with departmental guidelines
   * Given thrombosis prophylactic treatment in accordance with national guidelines

   Need for additional salvage thoracical surgery or non-surgical pleural procedures Following the primary intervention subsequent decisions during the admission to perform salvage thoracic surgery or additional non-surgical pleural procedures is made in accordance with the national guidelines from the Danish Society for Cardiothoracic Surgery and Danish Society for Respiratory Medicine.

   Removal of drain/pigtail

   The decision to remove the drain / pigtail is made by the clinician attending the patient. The following criteria are used as a guide for discontinuation of drain/pigtail in both groups:
   * Clinical improvement of the patient (e.g. no fever/subfebril, improved general condition)
   * Satisfactory biochemical response (with respect to a decrease in leukocytes and CRPs)
   * Imaging (TUS, CT or Chest X-ray (CXR) in 2 planes) without significant residual effusion (< 100 ml)
   * Drain with clear pleural fluid by rinsing In both groups removal of drain / pigtail does not await the results of any of the obtained cultures of the pleural fluid. As such the presence of negative cultures is used as removal criteria.

   Discharge from hospital

   In current usual practice in Denmark, patients with pleural empyema are typically discharged when:
   * The drain / pigtail has been removed
   * Antibiotic treatment has been changed from intravenous to oral treatment without signs of subsequent clinical or paraclinical treatment within one day following the change These principles are also used in the study.

   Data recording

   Prior to informed consent obtained as part of screening for study participation:
   * Data needed to determine whether inclusion criteria are met (see above)
   * Data needed to determine whether any exclusion criteria are present (see above)

   Baseline patient data: age, gender, comorbidities, medication, performance status, previously recorded lung function etc.

   Surgical and TUS data: used time, specific type of procedure, operator, drain size, complications etc.

   Drain data: Length of drain treatment, daily output / input, removal criteria, no. of drains used etc.

   Costs during hospitalization:

   Calculated for the two groups regarding the following expenses:
   * VATS Group:

     * Utensils used during surgery
     * Time of the procedure
     * Consumption of staff resources
     * Hospitalization time
     * Medicine
   * Drain group:

     * Equipment used during the procedure
     * Procedure Time
     * Consumption of human/staff resources
     * Fibrinolyticum and DNase (amount used)
     * Hospitalization time
     * Medicine

   Costs within the 1st year after discharge:

   Calculated for the two groups regarding the following expenses:
   * Re-admission
   * Ambulatory services
   * Medication
   * Number of sick days
   * Visit to a GP

   Patient satisfaction and functional level:

   • Data in the form of EQ5D and St. George Research Questionnaire is collected at the following times:
   * Upon inclusion in the study
   * At discharge
   * Outpatient data: 1, 3, 6 and 12 months.

   Various parameters acquired from and after hospitalization (including ambulant outpatient visits):
   * Hospitalization time, total and after commencement of intervention
   * Primary intervention considered as final treatment
   * In hospital and 30 day mortality
   * Drainage time
   * Radiological regression a.m. MIST II
   * Number and types of drains
   * Need for additional surgery during and within 12 months after hospitalization
   * Need for additional intrapleural therapy during and within 12 months after hospitalization
   * Need for intensive care therapy
   * Consumption of painkillers during hospitalization and within 12 months after hospitalization
   * Lung function tests and walking tests
   * Re-admission
   * Miscellaneous paraclinical parameters (e.g. biochemistry, microbiolology, pathology)

   Data obtained from National Patient Register:
   * Health related costs and expenses (e.g. hospital admissions, outpatient visits, general practice consultations, use of physiotherapy)
   * Prescribed medication
   * Death (e.g. date, cause)

   Outpatient follow-up after discharge In conjunction with participation in the project, in addition to any common local controls, outpatient follow-up is performed at the regional respiratory medicine out-patient-clinic after 3, 6 and 12 months after discharge.

   Data collection Media
   * REDCap (Research Electronic Data Capture), REDCap Consortium, Vanderbilt University Medical Center, Tennessee, USA
   * Electronic patient record (EPJ in Region Midt, EPJ in Region North, EPJ (COSMIC) in Region South and EPJ (EPIC Health Platform) in the Capital Region and Region Zealand).
   * Health related costs are retrieved via the National Patient Register (LPR).

   Handling and archiving data All data is entered in a Case Report Form in RedCap. REDCap is a professional database that provides a user-friendly interface. The REDCap data management system is secure, fully compliant with all regulatory guidelines, and includes a complete audit-trail for data entry validation. Through these mechanisms, as well as relevant training for all involved parties, patient confidentiality will be safeguarded. REDCap is available for free at both Odense and Aarhus University.

   When handling, processing and archiving data collected, the Data Inspectorate's guidelines are followed, which implies that all personal data are deleted at the end of the project. The collected data is stored at the Department of CardioThoracic and Vascular Surgery, Aarhus University Hospital and at Department of Pulmonology, Odense University Hospital.

   Sample size and power calculation The study is based on assumptions and knowledge about admission time, both from national and international publications. We calculated the sample size based on the following assumptions: the main effect target is the difference between the total time (primary endpoint) between the two groups of patients (VATS versus drainage). The distribution of the hospitalization time is expected to be skewed to the right, so that a logarithmic transformation is needed to achieve normality.

   We assume a median hospitalization period in the drainage group of 12 days, a minimum clinically relevant difference in hospitalization of two days, 80% power, and coefficient of variation (CV) of 40%.

   Significance level is set to 0.05. Thus, 77 patients in each group must be included. To account for excluded patients (set at 20%), we expect to include 92 patients in each group. A total of 184 patients is to be included.

   In terms of showing clinically relevant non-inferiority with a difference in hospitalization of 1 day with a 80% power, and CV of 40%, 70 patients is needed in each group. This is based on a true improvement of 1 hospitalization day. Based on the annual number of patients diagnosed with pleura empyema in Denmark, we find it feasible to include the needed number of patients in the trial during the inclusion period.

   Data analysis Data extractions are made from RedCap database. Data analysis is performed using one of the following: Microsoft® Excel® 2011 (Microsoft Corporation, Washington, USA), Prism Version 8 for Mac OS X (GraphPad Software, Inc., California, USA), STATA version 16 (StataCorp LLC, Texas, USA). Endpoints will be described for the individual group by median and percentile, assuming data is not normally distributed.

   Differences between the groups in the primary endpoint are determined by t-test at the log-entry time and reported as median ratios with associated confidence intervals. Patients dying during the admission is omitted from the analysis if the primary endpoint. Whether death before discharge affects the primary endpoint is assessed using survival analysis as sensitivity analysis. We expect that the distribution between stages II and III will be 75% and 25%, respectively, and whether there is a difference between stages II and III will be assessed as secondary analysis. When repeating measurements (e.g. quality of life), repeated measurements ANOVA are used with treatment and time as systematic effects and patient as random effect. All data are analyzed primarily according to the intention to treat principle, but there will also be one per protocol analysis regarding the above-mentioned endpoints. Comparison will take place between the two groups (drainage and VATS).

   Statistical cooperation partner Bo Martin Bibby. Ass. Professor, Biostatistical Advisory Service (BIAS), Faculty of Health Sciences, Aarhus University.

   Risks of participation, ethical considerations and monitoring Common clinical practice is currently very divergent and there is no national or international consensus on which of the treatments is preferable (VATS versus drainage). There is thus no safe evidence for any of the regimes.The individual patient may not immediately benefit from participating. The results of the study will primarily benefit future patients.

   Ethics and dissemination All patients provide informed consent before randomisation. The research project is carried out in accordance with the Helsinki II Declaration, European regulations and Good Clinical Practice Guidelines. The Scientific Ethics Committees for Denmark and the Danish Data Protection Agency have provided permission. Information about the subjects is protected under the Personal Data Processing Act and the Health Act. The trial is registered at www.clinicaltrials.gov, and monitored by the regional Good Clinical Practice monitoring unit. The results of this study will be published in peer-reviewed journals and presented at various national and international conferences.

   Interruption of the experiment Suspected Severe Adverse Reactions suspend the attempt for the individual patient. However, patient data is still used in the project according to intention to treat principles.

   Earlier termination of the trial for the individual patient
   * If the patient wishes to leave the study.
   * If unexpected complications occur If leaving the trial, the patient will follow the department's usual procedure for treating patients treated for pleura empyema. If the patient wishes to leave the study, the collected data is not used if, as a result of unexpected complications, the patient cannot receive the intervention the patient is randomized, the patient enters the data and continues to collect data in accordance with the intention to treat principles.

   Events and side effects All unintended events and adverse events throughout the treatment period and until the last call after 30 days are recorded. All Adverse Events are recorded in the patients Case Report Form.

   Agreements with other departments / hospitals All involved departments have signed a document obligating them to take active part in the trial.

   All Pulmonary and Thoracic Surgical departements on the four University Hospital has agreed to participate in the trial The Danish Society of Cardiothoracic Surgery and the Danish Society of Respiratory Medicine has both recommended and endorsed the study

   Project collaboration and work distribution The main applicant will be the principal investigator, and primarily responsible for the overall practical feasibility, conducting and hosting of the study. The co-applicants (Morten Bendixen and Thomas Decker Christensen) is part of the steering committee and equally responsible for the conduction of the trial.

   Morten Bendixen have taking part in the process of preparing and writing the protocol, organizing the study and applying for economical support. He will take part in the implementing of the study (inclusion of patients, performing surgery, practical issues etc.), analyzing and interpretation of data and writing of the manuscripts. His share of the budget is estimated to 1269400 Dkr.

   Thomas Decker Christensen have taking part in the idea/concept of the study, the process of preparing and writing the protocol, organizing the study and applying for economical support. He will take part in the implementing of the study (inclusion of patients, performing surgery, practical issues etc.), analyzing and interpretation of data and reviewing the manuscripts. His share of the budget is estimated to 1269400 Dkr.

   International collaborators

   To provide scientific input and an international perspective, we have assembled a group of international experts with great expertise and experience within pleural emphyema and clinical trials. This group include:
   * Prof. Najib. N. Rahman, Professor, Consultant of Respiratory Medicine, Nuffield Department of Medicine, Clinical Director, Oxford Respiratory Trials Unit, University of Oxford, UK
   * Eihab Bedawi, MD, Nuffield Department of Medicine, Clinical Director, Oxford Respiratory Trials Unit, University of Oxford, UK
   * Prof. Babu Naidu, Professor, Consultant of Thoracic Surgery, Department of Thoracic Surgery, Queen Elizabeth Hospital Birmingham, UK & Institute of Inflammation and Ageing, University of Birmingham, UK.

   Report / applied for permission from the following institutions
   * Scientific ethics committee
   * Data Inspectorate / Region Midt
   * Medicines Agency (Case No. 2017084202)
   * www.clinicaltrials.gov

   Time schedule The proposal covers a 5 years' timeline, with approximately half a year for further planning and organization of the trial, 2.5 years for patient inclusion, 1 year for follow-up and 1 year for data analyses and publications. Additional details are provided in the attached figure.

   Publications and sharing of the data Both positive, negative and inconclusive results from the study will be published in international journals. The researchers' free right to publication cannot be restricted. All information will be disclosed in anonymous form. The results will also be presented at international scientific congresses.

   A minimum of six manuscripts are planned from the current trial. Study findings will be published irrespective of the results. Completely de-identified data will be shared in public database after the trial to allow for other researchers to replicate the results or to test new hypotheses.

   Steering committee A steering committee will be responsible for the design and conduct of the trial. The principal investigator will be Christian B Laursen (see applicant information) Additional members of the multidisciplinary steering committee will include Thomas Decker Christensen (co-applicant), Morten Bendixen (co-applicant), Peter B. Licht MD, PhD (thoracic surgery), Rene H. Petersen MD, PhD (thoracic surgery), Lars Møller MD (thoracic surgery), Jens-Ulrik Stæhr Jensen MD, PhD (pulmonologist), Vasiliki Panou MD (pulmonologist) and Søren Helbo Skaarup MD (pulmonologist).

   A qualified Ph.D. fellow will be included in the steering committee and involved in the conduct of the trial.

   Abbreviations used in the project description CRP: C-reactive protein CT: Computed tomography CXR:Chest X-ray EQ5D: European Quality of Life F: French Ml: Milliliter MIST: Multi-centre Intra-pleural Sepsis Trial TUS: Thoracic Ultrasound ULS: Ultrasound VATS: Video Assisted Thoracoscopic Surgery

ELIGIBILITY:
Inclusion Criteria:

* 18 years or more on the day of hospitalization
* Must be able to provide informed consent
* Acute hospitalization within the last 48 hours
* Meeting diagnostic criteria for community acquired pleural infection using the following criteria:

  1. A clinical presentation compatible with pleural infection AND
  2. Has pleural fluid which is either:

     1. purulent pleural fluid or
     2. gram stain positive or
     3. culture positive or
     4. acidic with pH < 7.2 or
     5. low pleural fluid glucose (< 2 mmol/L) in the absence of accurate pH measurement or
     6. septated pleural fluid on ultrasound

Exclusion Criteria:

* • Pregnancy. Prior to inclusion of fertile women (defined as the period from menarche to postmenopause) a negative pregnancy test must be available
* Breastfeeding
* Declared terminally ill or a predicted survival of less than 3 months
* Previous intrathoracic surgery (within <1 year on the same side of the thorax as where the parapneumonic effusion/pleural empyema is located
* Previously (within <1 year) hospitalized with with complex parapneumonic effusion (stage II) or pleural empyema (stage III)
* Drainage during the current admission on the same side of the thorax (excluding diagnostic pleural puncture)
* Hospitalization within 7 days prior to current hospitalization
* Previous allergic reaction to alteplase or DNase
* Use of alteplase therapy contraindicated:

  * Ongoing treatment with oral anticoagulant incl. new oral anticoagulants (e.g. warfarin (Marevan), Dabigatranetexilat (Pradaxa), Rivaroxaban (Xarelto), Apixaban (Eliquis), Endoxaban (Lixiana))
  * Significant ongoing bleeding or within last six months
  * Known haemorrhagic diathesis
  * Previous or suspected intracranial hemorrhage
  * Suspected subarachnoidal hemorrhage or condition following subarachnoidal hemorrhage from aneurysm
  * All forms of damage to the central nervous system (e.g. cerebral tumors, aneurysm, intracranial / spinal surgery)
  * Recent (within 10 days) cardiac resuscitation, birth, or perforation of non-compressible blood vessel (e.g. puncture of v. subclavia, v. jugularis)
  * Severe, uncontrolled arterial hypertension
  * Bacterial endocarditis, pericarditis
  * Acute pancreatitis
  * Documented ulcerative gastrointestinal disease within last 3 months, esophagal varices, arterial aneurysm, arterio-venous malformations
  * Tumor / malignancy with an increased risk of hemorrhage
  * Severe liver disease, including liver failure cirrhosis, portal hypertension (esophagal varices), and active hepatitis
  * Large operation or significant trauma within previous 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2022-10-30 (Actual); Primary Completion 2027-10-30 (Estimated); Study Completion 2028-10-30 (Estimated)

PRIMARY OUTCOMES:
Length of hospital stay | Through study completion, an average of 1 year
  Admission time is defined as the time from first admission in the course of the hospitalization and to the completion of treatment defined as time of discharge from hospital without need of any additional invasive treatment.

SECONDARY OUTCOMES:
Length of hospital stay in subgroups | Through study completion, an average of 1 year
  patients are stratified in subgroups (Stage, TUS score, RAPID score)
Length of hospital stay after commencement of intervention | Through study completion, an average of 1 year
  Length of hospital stay after the time for starting the intervention
Days at home up to 30 days after intervention (DAH30) treatment | Through study completion, an average of 1 year
  Days at home up to 30 days after intervention (DAH30) treatment
30-day and in-hospital mortality | Through study completion, an average of 1 year
  30-day and in-hospital mortality
Proportion of patients where primary intervention could be considered as definitive treatment | 30 days
  Proportion of patients where primary intervention could be considered as definitive treatment
Complications ranked by Clavien-Dindo classification and Comprehensive Complication Index (CCI) | Through study completion, an average of 1 year
  Complications ranked by Clavien-Dindo classification and Comprehensive Complication Index (CCI)
Need for additional thoracic surgery within 12 months after hospitalization | 1 year
  Need for additional thoracic surgery within 12 months after hospitalization
Consumption of painkillers during hospitalization and within 12 months after hospitalization | Through study completion, an average of 1 year
  Consumption of painkillers during hospitalization and within 12 months after hospitalization
Lung physiology within 12 months after hospitalization | 1 year
  Lung physiology within 12 months after hospitalization
Quality of life and patient reported outcomes within 12 months after hospitalization | Through study completion, an average of 1 year
  Quality of life and patient reported outcomes within 12 months after hospitalization (measured by European Quality of life (EQ5D)) EQ-5D is a generic quality of life questionnaire that comprises five questions, each with three possible answers. The five questions refer to various dimensions of health-related quality of life: mobility, self-care, usual activities, pain, and anxiety/depression, respectively. Each question is answered with either "no problems", "some problems", or "severe problems"
Health related costs | 1 year
  Health related costs within 12 months after hospitalization hospitalization.The unit is in Euro's).
  Costs were defined as use of any resource item multiplied by a unit cost. We used a marginal cost concept. That is, we limited the cost measurement to resource items that differed between the two procedures whereas costs that were unaffected by treatment procedure were not included in the analysis. The latter included administrative costs, buildings, electricity, heating, and water.
  For each patient, we calculated the cost of surgery and drainage, inpatient hospital stays and outpatient hospital visits, consultations with general practitioners, and use of prescription drugs during 52 weeks following intervention.
  Information on the use of healthcare after discharge was collected from the Danish National Patient Register, The National Health Service Register and The Danish National Prescription Registry, all administered by Statistics Denmark.
Quality of life and patient reported outcomes within 12 months after hospitalization | Through study completion, an average of 1 year
  Quality of life and patient reported outcomes within 12 months after hospitalization (measured by St. George Research Questionnaire) St. George Research Questionnaire (respiratory) consist of 14 questions which can be answered either True or False.

CONTACTS AND LOCATIONS:
Overall Officials: Christian B Laursen, MD, PhD, Principal Investigator — Odense University Hospital; Christian B Laursen, MD, PhD, Principal Investigator — Department of Respiratory Medicine, Odense University Hospital, Odense, Denmark
Locations (3):
- Denmark (3):
  - Aarhus University Hospital, Aarhus, Aarhus
  - Rigshospitalet, Copenhagen
  - Odense University Hospital, Odense

IPD SHARING:
Plan to Share IPD: Yes
All data can be shared , but the data will not be person attributable, so the individual patient can not be identified
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After completion of the study - after / during the publication process
Access Criteria: Mail to the principle investigator

REFERENCES:
- [Background] Maskell NA, Davies CW, Nunn AJ, Hedley EL, Gleeson FV, Miller R, Gabe R, Rees GL, Peto TE, Woodhead MA, Lane DJ, Darbyshire JH, Davies RJ; First Multicenter Intrapleural Sepsis Trial (MIST1) Group. U.K. Controlled trial of intrapleural streptokinase for pleural infection. N Engl J Med. 2005 Mar 3;352(9):865-74. doi: 10.1056/NEJMoa042473. PMID 15745977
- [Background] Davies HE, Davies RJ, Davies CW; BTS Pleural Disease Guideline Group. Management of pleural infection in adults: British Thoracic Society Pleural Disease Guideline 2010. Thorax. 2010 Aug;65 Suppl 2:ii41-53. doi: 10.1136/thx.2010.137000. No abstract available. PMID 20696693
- [Background] Molnar TF. Current surgical treatment of thoracic empyema in adults. Eur J Cardiothorac Surg. 2007 Sep;32(3):422-30. doi: 10.1016/j.ejcts.2007.05.028. Epub 2007 Jul 23. PMID 17646107
- [Background] Tokuda Y, Matsushima D, Stein GH, Miyagi S. Intrapleural fibrinolytic agents for empyema and complicated parapneumonic effusions: a meta-analysis. Chest. 2006 Mar;129(3):783-90. doi: 10.1378/chest.129.3.783. PMID 16537882
- [Background] Hooper CE, Edey AJ, Wallis A, Clive AO, Morley A, White P, Medford AR, Harvey JE, Darby M, Zahan-Evans N, Maskell NA. Pleural irrigation trial (PIT): a randomised controlled trial of pleural irrigation with normal saline versus standard care in patients with pleural infection. Eur Respir J. 2015 Aug;46(2):456-63. doi: 10.1183/09031936.00147214. Epub 2015 May 28. PMID 26022948
- [Background] Rahman NM, Maskell NA, West A, Teoh R, Arnold A, Mackinlay C, Peckham D, Davies CW, Ali N, Kinnear W, Bentley A, Kahan BC, Wrightson JM, Davies HE, Hooper CE, Lee YC, Hedley EL, Crosthwaite N, Choo L, Helm EJ, Gleeson FV, Nunn AJ, Davies RJ. Intrapleural use of tissue plasminogen activator and DNase in pleural infection. N Engl J Med. 2011 Aug 11;365(6):518-26. doi: 10.1056/NEJMoa1012740. PMID 21830966
- [Background] Scarci M, Abah U, Solli P, Page A, Waller D, van Schil P, Melfi F, Schmid RA, Athanassiadi K, Sousa Uva M, Cardillo G. EACTS expert consensus statement for surgical management of pleural empyema. Eur J Cardiothorac Surg. 2015 Nov;48(5):642-53. doi: 10.1093/ejcts/ezv272. Epub 2015 Aug 7. PMID 26254467
- [Background] Bagheri R, Tavassoli A, Haghi SZ, Attaran D, Sadrizadeh A, Asnaashari A, Basiri R, Salehi M, Moghadam KA, Tabari A, Sheibani S. The role of thoracoscopic debridement in the treatment of parapneumonic empyema. Asian Cardiovasc Thorac Ann. 2013 Aug;21(4):443-6. doi: 10.1177/0218492312466858. Epub 2013 Jul 11. PMID 24570527
- [Background] Redden MD, Chin TY, van Driel ML. Surgical versus non-surgical management for pleural empyema. Cochrane Database Syst Rev. 2017 Mar 17;3(3):CD010651. doi: 10.1002/14651858.CD010651.pub2. PMID 28304084
- [Background] Koppurapu V, Meena N. A review of the management of complex para-pneumonic effusion in adults. J Thorac Dis. 2017 Jul;9(7):2135-2141. doi: 10.21037/jtd.2017.06.21. PMID 28840015
- [Background] Bishay M, Short M, Shah K, Nagraj S, Arul S, Parikh D, Jawaheer G. Efficacy of video-assisted thoracoscopic surgery in managing childhood empyema: a large single-centre study. J Pediatr Surg. 2009 Feb;44(2):337-42. doi: 10.1016/j.jpedsurg.2008.10.083. PMID 19231530
- [Background] Ravn, J. Should all patients with pleural emphyema be referred to a thoracic operation? Dan. Med. J. 179, V69273 (2017).
- [Background] Psallidas I, Yousuf A, Talwar A, Hallifax RJ, Mishra EK, Corcoran JP, Ali N, Rahman NM. Assessment of patient-reported outcome measures in pleural interventions. BMJ Open Respir Res. 2017 Jul 3;4(1):e000171. doi: 10.1136/bmjresp-2016-000171. eCollection 2017. PMID 28883922
- [Background] Rahman NM, Kahan BC, Miller RF, Gleeson FV, Nunn AJ, Maskell NA. A clinical score (RAPID) to identify those at risk for poor outcome at presentation in patients with pleural infection. Chest. 2014 Apr;145(4):848-855. doi: 10.1378/chest.13-1558. PMID 24264558
- [Derived] Christensen TD, Bendixen M, Skaarup SH, Jensen JU, Petersen RH, Christensen M, Licht P, Neckelmann K, Bibby BM, Moller LB, Bodtger U, Borg MH, Saghir Z, Langfeldt S, Harders SMW, Bedawi EO, Naidu B, Rahman N, Laursen CB. Intrapleural fibrinolysis and DNase versus video-assisted thoracic surgery (VATS) for the treatment of pleural empyema (FIVERVATS): protocol for a randomised, controlled trial - surgery as first-line treatment. BMJ Open. 2022 Mar 9;12(3):e054236. doi: 10.1136/bmjopen-2021-054236. PMID 35264347